CLINICAL TRIAL: NCT04162067
Title: Type 1 Diabetes in Canada: The Demographic, Care Profiles and Glycemic Control of Patients Living With Type 1 Diabetes From the LMC Diabetes Patient Registry
Brief Title: The Current Health Status of Patients Living With Type 1 Diabetes From the LMC Diabetes Patient Registry
Status: Completed | Type: Observational
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: T1D Registry
Record Dates: First submitted 2019-11-10; First posted 2019-11-14 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Type1diabetes
Keywords: Diabetes Mellitus, Type 1; hypoglycemia; hemoglobin A1c; time in range; continuous glucose monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study uses the Canadian LMC Diabetes Registry to describe the current health status of Canadians with type 1 diabetes. The study provides a detailed report of the demographic composition, treatment regimens, self-care approaches, health status, metabolic outcomes, and glycemic control of a large Canadian community-based, specialist-led cohort of patients with type 1 diabetes. Specific study outcomes will also be evaluated in a subgroup of patients using continuous subcutaneous insulin infusion (CSII) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes for ≥ 6 months
* Assessed by an LMC endocrinologist between July 1, 2015 and June 30, 2018
* Followed by an LMC endocrinologist for > 6 months
* Informed consent provided and signed for medical record data to be used for research purposes

Exclusion Criteria:

* clinical diagnosis of type 2 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 diabetes under the care of an endocrinologist at an LMC Healthcare centre, in the provinces of Ontario, Quebec, or Alberta, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
HbA1c | 1 day
  HbA1c will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019

SECONDARY OUTCOMES:
Fasting plasma glucose | 1 day
  Fasting plasma glucose will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019
Proportion of patients with HbA1c ≤7.0%, 7.1 to 8.0%, 8.1 to 9.0% and >9.0% | 1 day
  HbA1c will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019
Lipid parameters | 1 day
  Mean LDL cholesterol (mmol/L), mean HDL cholesterol (mmol/L), mean non-HDL cholesterol (mmol/L) and mean triglycerides (mmol/L) will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019
Proportion of patients below and above target LDL cholesterol | 1 day
  LDL cholesterol (mmol/L) will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019
Blood pressure | 1 day
  Mean systolic blood pressure (mmHg) and mean diastolic blood pressure (mmHg) will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019
estimated glomerular filtration rate (eGFR) | 1 day
  Proportion of patients (%) with eGFR <30 mL/min/1.73 m2, between 30-60 mL/min/1.73 m2, and >60 mL/min/1.73 m2 will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019
Albuminuria | 1 day
  Proportion of patients (%) with urine albumin to creatinine ratio (uACR) <2.0 mg/mmol and ≥ 2.0 mg/mmol will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019
Weight | 1 day
  Mean body weight (kg) will be measured by accessing patients medical records and it will be evaluated at one time point only.The value will be the last measured value for each patient between January 2015 and June 2019
Body mass index (BMI) | 1 day
  Mean BMI (kg/m2) and proportion of patients (%) with BMI <18.5, 18.5 to <25, 25 to <30 and ≥ 30 kg/m2, will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019.
Waist circumference | 1 day
  Mean waist circumference (cm) will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019
Thyroid stimulating hormone (TSH) | 1 day
  Mean thyroid stimulating hormone (µIU/mL) will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019
Alanine aminotransferase (ALT) | 1 day
  Mean ALT (U) will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019
Microvascular comorbidity | 1 day
  History of any of the following: retinopathy, neuropathy or nephropathy. The history will be accessed from the patients medical records.
Macrovascular comorbidity | 1 day
  History of any of the following: coronary artery disease, angina, cardiovascular disease, congestive heart failure, coronary vascular disease, myocardial infarction, coronary artery bypass grafting, angioplasty, cerebral vascular disease, stroke, cerebrovascular accident, peripheral vascular disease, atherosclerotic disease, intermittent claudication, aorto-femoral bypass or femoral popliteal bypass. The history will be accessed from the patients medical records.
Weekly incidence of any hypoglycemia | 1 day
  Self-reported weekly incidence of any hypoglycemia will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019
Yearly incidence of severe hypoglycemia | 1 day
  Self-reported yearly incidence of hypoglycemia will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019
Mental health comorbidity | 1 day
  History of any of the following: anxiety, depression, bipolar affective disorder, eating disorder, schizophrenia, sleep disorder. The history will be accessed from the patients medical records.
Erectile dysfunction | 1 day
  Proportion of males with erectile dysfunction. The medical history will be accessed from the patients medical records.
Insulin type | 1 day
  Proportion of patients (%) using rapid-acting, intermediate acting and long-acting insulin
Insulin therapy regimen | 1 day
  Proportion of patients (%) using multiple daily injections (MDI) and continuous subcutaneous insulin infusion (CSII)
Pump model | 1 day
  Proportion of patients (%) using different types of pump models.
Adjunct diabetes therapies | 1 day
  Proportion of patients (%) using non-insulin diabetes therapies, including metformin, SGLT2 inhibitors, DPP4 inhibitors, and GLP-1 receptor agonists
Lipid lowering therapies | 1 day
  Proportion of patients (%) using lipid lowering therapies
Antihypertensive therapies | 1 day
  Proportion of patients (%) using antihypertensive therapies
Mental health therapies | 1 day
  Proportion of patients (%) using therapies for a mental health condition
Glucose meter use | 1 day
  Proportion of patients (%) using a blood glucose monitor
Continuous glucose monitor (CGM) use | 1 day
  Proportion of patients (%) using a CGM device or a flash glucose monitor device
Glucagon availability | 1 day
  Proportion of patients (%) using glucagon
Clinical outcomes stratified by age group | 1 day
  Age groups include 18-25 years, 26-49 years, and greater or equal to 50 years

OTHER OUTCOMES:
Mean CGM glucose | 5 to 90 days
  Mean CGM glucose in sub-group of patients with available CGM data. The last 5 to 90 days of the patients CGM data will be accessed from the patients medical records.
Time in range | 5 to 90 days
  Percentage of time with CGM glucose concentration between 4-10 mmol/L in sub-group of patients with available CGM data. The last 5 to 90 days of the patients CGM data will be accessed from the patients medical records.
Time in hypoglycemia | 5 to 90 days
  Percentage of time with CGM glucose concentration < 4 mmol/L in sub-group of patients with available CGM data. The last 5 to 90 days of the patients CGM data will be accessed from the patients medical records.
Time in hyperglycemia | 5 to 90 days
  Percentage of time with CGM glucose concentration > 10 mmol/L in sub-group of patients with available CGM data. The last 5 to 90 days of the patients CGM data will be accessed from the patients medical records.
Standard deviation (SD) of CGM glucose | 5 to 90 days
  SD (mmol/L) of CGM glucose in sub-group of patients with available CGM data. The last 5 to 90 days of the patients CGM data will be accessed from the patients medical records.
Co-efficient of variation (CV) of CGM glucose | 5 to 90 days
  Proportion of patients with CV ≤ 36% and CV >36% in sub-group of patients with available CGM data. The last 5 to 90 days of the patients CGM data will be accessed from the patients medical records.
HbA1c at referral | 1 day
  Mean HbA1c (%) in the six months prior to referral. The last measured value will be used and will be accessed through the patients medical records.
HbA1c in sub-group of patients using CSII therapy | 1 day
  HbA1c will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019.
Brand of insulin pump | 1 day
  The proportion of patients using each type of insulin pump model will be reported in the sub-group of patients using CSII therapy
Brand of bolus insulin | 1 day
  The proportion of patients using each type of bolus insulin brand will be reported in the sub-group of patients using CSII therapy
Sociodemographics in the subgroup of patients using CSII therapy | 1 day
  Sociodemographics include age, gender, ethnicity, education, household income and health coverage.
Weekly incidence of any self-reported hypoglcyemia in the subgroup of patients using CSII therapy | 1 day
  Weekly incidence of any self-reported hypoglycemia will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019.
Yearly incidence of severe hypoglycemia in the subgroup of patients using CSII therapy | 1 day
  Yearly incidence of severe hypoglycemia will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019.
Weight in the subgroup of patients using CSII therapy | 1 day
  Weight will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019.
BMI in the subgroup of patients using CSII therapy | 1 day
  BMI will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019.
eGFR in the subgroup of patients using CSII therapy | 1 day
  eGFR will be expressed as the proportion of patients with eGFR <30, 30 to 60 and >60 mL/min/1.73 m2. eGFR will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019.
LDL-cholesterol in the subgroup of patients using CSII therapy | 1 day
  LDL cholesterol will be expressed as a mean and the proportion of patients with LDL-cholesterol ≤ 2 mmol/L and >2 mmol/L. LDL cholesterol will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019.
Blood pressure in the subgroup of patients using CSII therapy | 1 day
  Blood pressure will be measured by accessing patients medical records and it will be evaluated at one time point only. The value will be the last measured value for each patient between January 2015 and June 2019.
Comorbidities in the subgroup of patients using CSII therapy | 1 day
  Comorbidities include microvascular complications and macrovascular complications.
HbA1c in the subgroup of patients using CSII therapy and using a do-it-yourself (DIY) closed loop system | 1 day
  The last available HbA1c measurement will be used that was collected between January 2015 and June 2019
HbA1c in the subgroup of patients using CSII therapy and using a hybrid closed loop system | 1 day
  The last available HbA1c measurement will be used that was collected between January 2015 and June 2019
HbA1c in the subgroup of patients using CSII therapy, stratified by age group | 1 day
  The last available HbA1c measurement will be used that was collected between January 2015 and June 2019. Age categories will include 18-25 years, 26-49 years, and greater than or equal to 50 years.
CGM metrics in the subgroup of patients using CSII therapy and a CGM device | 5 to 90 days
  CGM metrics include: mean CGM glucose, SD of CGM glucose, time in range, time in hyperglycemia, time in hypoglycemia, and co-efficient of variation of CGM glucose. The last 5 to 90 days of patients data will be used.
HbA1c in the subgroup of patients using a CGM device | 1 day
  The last available HbA1c measurement will be used that was collected between January 2015 and June 2019. This outcome will be further stratified by CSII vs MDI therapy.
HbA1c in the subgroup of patients using CSII therapy, stratified by mean self-measured blood glucose testing frequency. | one week
  HbA1c will be evaluated in patients who have a mean daily testing frequency < two times/day and ≥ two times/day. The last week of recorded self-measured blood glucose testing frequency data will be used (between January 2015 and June 2019).
HbA1c in the subgroup of patients using CSII therapy, stratified by patients considered "atypical" for pumping by Canadian regulatory authorities | one week
  HbA1c will be evaluated in patients who use carbohydrate counting to calculate insulin dose <50% of the time and <20% of the time

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Aronson, MD, Principal Investigator — LMC Healthcare
Locations (1):
- LMC Healthcare, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aronson R, Brown RE, Abitbol A, Goldenberg R, Yared Z, Ajala B, Yale JF. The Canadian LMC Diabetes Registry: A Profile of the Demographics, Management, and Outcomes of Individuals with Type 1 Diabetes. Diabetes Technol Ther. 2021 Jan;23(1):31-40. doi: 10.1089/dia.2020.0204. Epub 2020 Jul 31. PMID 32667835